CLINICAL TRIAL: NCT06582862
Title: The Effect of Aerobic and Anaerobic Exercise
Brief Title: The Effect of Aerobic and Anaerobic Exercise on Oxidative Stress and Cellular Fitness in Healthy Trained Young Men
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Novi Silvia Hardiany, Research Coordinator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-05-0791
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Health, Subjective
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 2 groups. One group will do aerobic exercise and other group will do anaerobic exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre aerobic exercise treatment (Experimental): Subject will do aerobic exercise 3 times a week for 1 month. The training program includes the following: Week 1 consists of interval running (2 sets of 10 repetitions of 400 meters each) with 3 minutes of rest between repetitions and 10 minutes of rest between sets. Week 2 transitions to continuous running for 15-20 minutes. Week 3 involves 30 minutes of cross-country running. In Week 4, the program returns to interval running as in Week 1.
  Interventions: Other: Exercise
- Pre anaerobic exercise treatment (Experimental): Subject will do anerobic exercise 3 times a week for 1 month. The sprint training program includes the following: In Weeks 1 and 3, perform sprints of 20 m, 40 m, 60 m, and 80 m, with 2 sets of 5 repetitions each, allowing 5 minutes of rest between repetitions and 10 minutes of rest between sets. In Weeks 2 and 4, run 2 sets of 5 repetitions of 50 m sprints, with 5 minutes of rest between repetitions and 10 minutes between sets.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Subjects will do aerobic and anaerobic exercise

SUMMARY:
This study aims to analyze the effects of aerobic and anaerobic exercise on health at the molecular level. By examining these effects, the study seeks to provide the public with insights into which types of exercise offer the most significant health benefits. Participants will engage in aerobic and anaerobic exercises for one month, with 5 mL of venous blood collected by experienced phlebotomists both before and after the exercise period. While blood collection may cause mild discomfort and temporary bruising, these symptoms should subside within a few days. The collected blood will be processed to separate plasma and leukocytes for the assessment of oxidative damage, lipid profile and cellular fitness parameters. The oxidative damage markers to be measured include malondialdehyde (MDA) levels, H2O2, and antioxidants such as total antioxidant capacity, superoxide dismutase, and glutathione peroxidase. Cellular fitness will be evaluated by measuring mitochondrial biogenesis markers (succinate dehydrogenase and PGC-1A), ATP levels, and ATPase inhibitor levels. The benefits for the participants, they will receive include a laboratory assessment to evaluate cell damage, lipid profiles, and mitochondrial function. Additionally, the study results will help identify the most beneficial type of physical exercise for optimal health.

DETAILED DESCRIPTION:
Oxidative stress arises from an imbalance between pro-oxidant and antioxidant levels, where the pro-oxidant status, primarily reactive oxygen species (ROS), exceeds the antioxidant defense. This imbalance can damage cellular components such as membranes, lipids, proteins, DNA, and lipoproteins, leading to various chronic and degenerative diseases. The human body defends against oxidative stress through antioxidant mechanisms. Numerous studies have shown that physical exercise increases ROS production, mainly through enhanced activity of phospholipase A2 (PLA2), nicotinamide adenine dinucleotide phosphate (NADPH) oxidase, and xanthine oxidase (XO). If ROS accumulates excessively, it can result in oxidative stress. During anaerobic exercise, lipid peroxidation levels can rise significantly for up to 48 hours post-exercise. The primary sources of free radical production during exercise include the mitochondrial electron transport chain, ischemia-reperfusion injury, and local inflammation, all of which induce oxidative stress.

Acute changes in oxidative stress biomarkers after exercise are often accompanied by an increase in antioxidant response. For instance, levels of uric acid (UA), catalase (CAT), and glutathione peroxidase (GPX) increase after 10 minutes to 4-8 hours of anaerobic exercise. Various types of exercise also stimulate mitochondrial biogenesis, though it remains unclear whether anaerobic or aerobic exercise is more effective in promoting this process in humans. Mitochondria, critical for cellular energy production, generate energy by transferring electrons from food into the respiratory chain system, involving various complex proteins. High-intensity interval training (HIIT) in aerobic exercises like cycling and walking prompts cells to produce more proteins for mitochondria and their ribosomes, effectively counteracting cellular aging. Endurance exercise (low to moderate intensity for 30 to 60 minutes) is well-known to enhance mitochondrial function in skeletal muscle, though the effects of anaerobic exercise on mitochondrial biogenesis are less studied.

Both aerobic and anaerobic exercises positively affect lipid metabolism. Aerobic exercise is particularly effective in improving lipid profiles, notably increasing high-density lipoprotein (HDL). An Australian study showed that aerobic exercise significantly reduced total cholesterol, low-density lipoprotein (LDL), and triglycerides (TG), while increasing HDL by about 0.05 mmol/L. A meta-analysis by Kelley et al. concluded that aerobic exercise increases HDL by 9% and reduces TG by 11%, though it does not significantly alter total cholesterol or LDL levels. Anaerobic exercise has also shown positive effects on lipid profiles. A European study on 16 obese subjects found that combined aerobic and anaerobic training led to a greater reduction in non-esterified fatty acids and body mass index than aerobic training alone.

In summary, physical exercise impacts oxidative stress, mitochondrial function, and metabolic parameters, yet the distinct effects of aerobic versus anaerobic exercise on these factors remain unclear. Aerobic and anaerobic exercises differ primarily in their oxygen (O2) requirements. Aerobic exercises, such as long-distance running, cycling, and jogging, are performed at low to moderate intensity (40% to 70% of VO2max) and rely on oxygen for sustained periods. Anaerobic exercise is performed at high intensity (75% to 100% of VO2 max) and does not rely on oxygen (O2) supply. Examples include sprints of 100 meters or less, throwing sports, and similar activities.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-23.
* body weight of 56-70 kg and a height of 158-175 cm.
* Systolic blood pressure values below 130 mmHg, and diastolic blood pressure below 90 mmHg.
* maximum oxygen consumption (VO2max) is calculated to be greater than 40 mL/(kg-minute).

Exclusion Criteria:

* fever
* having chronic diseases (heart disease, lung disease)
* smoking

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of Malondialdehyde (MDA) | 1 month
  MDA in nmoL/mL is measured using spectrophotometer from the subject's plasma
Concentration of Hydrogen Peroxide | 1 month
  Hydrogen peroxide in mmol/L is measured using spectrophotometer from the subject's plasma
Concentration of Superoxide dismutase (SOD) | 1 month
  SOD in U/mL is measured using spectrophotometer from the subject's plasma
Concentration of Total Antioxidant Capacity | 1 month
  Total Antioxidant Capacity in U/mL is measured using spectrophotometer from the subject's plasma
Concentration of Glutathione Peroxidase (GPx) | 1 month
  GPx in in U/mL is measured using spectrophotometer from the subject's plasma

SECONDARY OUTCOMES:
Concentration of Succinate Dehydrogenase (SDH) | 1 month
  SDH in U/L is measured using spectrophotometer from the peripheral blood mononuclear cells of subject
Concentration of Peroxisome proliferator-activated receptor-gamma coactivator (PGC)-1alpha | 1 month
  PGC-1alpha in ng/mL is measured using spectrophotometer from the the peripheral blood mononuclear cells of subject
Concentration of Adenosine triphosphate (ATP) | 1 month
  ATP in micromole/L is measured using spectrophotometer from the the peripheral blood mononuclear cells of subject
Concentration of ATPase inhibitor | 1 month
  ATPase inhibitor in ng/mL is measured using spectrophotometer from the the peripheral blood mononuclear cells of subject

CONTACTS AND LOCATIONS:
Overall Officials: Novi Hardiany, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No